CLINICAL TRIAL: NCT03445689
Title: Oxygenation Instability and Maturation of Control of Breathing in Premature Infants
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nelson Claure, Associate Professor, University of Miami
Other Study IDs: 20161114; U01HL133689 (NIH)
Record Dates: First submitted 2018-02-06; First posted 2018-02-26 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Infant,Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of oxygenation instability — Recordings of SpO2 and heart rate will be analyzed by dedicated software to obtain frequency, duration and severity of episodes of hypoxemia and hyperoxemia.
Other: Determination of mechanisms of hypoxemia episodes — Recordings of SpO2, heart rate, esophageal pressure, tidal volume, minute volume, respiratory rate and transcutaneous PCO2 will be analyzed to determine the prevalence, severity and duration of hypoxemia episodes produced by the different mechanisms.
Other: Assessment of respiratory instability — Recordings of tidal volume, minute volume and respiratory rate will be analyzed to determine frequency of apnea, periodic breathing, distribution of inter-breath intervals.
Other: apneic threshold of CO2 — In mechanically ventilated infants the apneic threshold of CO2 will be measured by transcutaneous PCO2 following a step wise increase in ventilator rate until spontaneous breathing ceases transiently. In spontaneously breathing infants the apnea threshold of CO2 will be measured during episodes central apnea.
Other: Assessment of peripheral chemoreceptor function — The Dejours test will be used to assess peripheral chemoreceptor function by measuring the immediate ventilatory response to high-inspired oxygen.
  Other Names: Dejours test
Other: Assessment of central chemo-receptor function — Central chemo-receptor function will be assessed by measuring the ventilatory response to inspired CO2.
  Other Names: Ventilatory response to CO2

SUMMARY:
Premature infants present with significant oxygenation instability in the form of frequent spontaneous episodes of hypoxemia during the first weeks after birth. These infants are also exposed to hyperoxemia.

The objective of this study is to determine the extent to which exposure to frequent episodes of hypoxemia and hyperoxemia in extreme premature infants during the early stages of their evolving lung disease is associated with altered maturation and function of their respiratory control system.

This study is part of the Prematurity-Related Ventilatory Control (Pre-Vent): Role in Respiratory Outcomes Clinical Research Centers (CRC) (U01) cooperative program of the National Heart Lung and Blood Institute (NHLBI) of the National Institutes of Health (NIH).

DETAILED DESCRIPTION:
Most extreme premature infants present with respiratory failure due to altered lung function compounded by breathing instability due to an immature respiratory control function.

Premature infants present with significant oxygenation instability in the form of frequent spontaneous episodes of hypoxemia during the first weeks after birth. As a result, these infants receive oxygen supplementation but this is often excessive and these infants are also exposed to hyperoxemia. The extent to which these episodes of hypoxemia or the exposure to hyperoxemia impact on the maturation and function of the control of breathing system in extreme premature infants during the evolving stages of their respiratory disease is unknown. This is a prospective study that will systematically evaluate such association in extreme premature infants.

The main objective of this study is to determine the extent to which exposure to frequent episodes of hypoxemia and hyperoxemia in extreme premature infants during the early stages of their evolving lung disease is associated with altered maturation and function of their respiratory control system.

This study is part of the Prematurity-Related Ventilatory Control (Pre-Vent): Role in Respiratory Outcomes Clinical Research Centers (CRC) (U01) cooperative program of the National Heart Lung and Blood Institute (NHLBI) of the National Institutes of Health (NIH).

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born at 23 0/7- 28 6/7 weeks gestational age
* Postnatal age up to equivalent to 36 weeks postmenstrual age
* Requiring supplemental oxygen and/or receiving mechanical ventilation, CPAP, nasal ventilation or nasal cannula

Exclusion Criteria:

* Severe congenital anomalies that may affect life expectancy or pulmonary or neurosensory development
* Severe CNS pathology that may alter respiratory control function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants admitted to the neonatal intensive care unit will be screened and will be considered eligible for inclusion if they fulfill all of the following inclusion and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Peripheral chemoreceptor control of breathing function | at 32 weeks corrected postmenstrual age
  Ventilatory response to oxygen (Dejours test)
Peripheral chemoreceptor control of breathing function | at 36 weeks corrected postmenstrual age
  Ventilatory response to oxygen (Dejours test)
Central chemoreceptor control of breathing function | at 32 weeks corrected postmenstrual age
  Ventilatory response to carbon dioxide
Central chemoreceptor control of breathing function | at 36 weeks corrected postmenstrual age
  Ventilatory response to carbon dioxide
Change in peripheral chemoreceptor control of breathing function | Change from 32 to 36 weeks postmenstrual age
  Ventilatory response to oxygen (Dejours test)
Change in central chemoreceptor control of breathing function | Change from 32 to 36 weeks postmenstrual age
  Ventilatory response to carbon dioxide

SECONDARY OUTCOMES:
Ventilatory stability - Apnea frequency | at 32 and 36 weeks corrected postmenstrual age
  Frequency of apnea episodes per hour
Ventilatory stability - Periodic breathing density | at 32 and 36 weeks corrected postmenstrual age
  Percent of time with periodic breathing
Ventilatory stability - Time series analysis of inter-breath interval | at 32 and 36 weeks corrected postmenstrual age
  Tail slope of the log-scaled probability density function of the inter-breath time series
Mechanisms of episodic hypoxemia | at 32 and 36 weeks corrected postmenstrual age
  Classify etiology of episodes of hypoxemia as central, obstructive, or mixed apnea or active exhalation based on measurements of respiratory inductance plethysmography, esophageal pressure
Apneic CO2 threshold in central apnea | at 32 and 36 weeks corrected postmenstrual age
  Carbon dioxide level change at onset of central apnea
Apneic CO2 threshold during mechanical ventilation | at 32 and 36 weeks corrected postmenstrual age
  Carbon dioxide level change at onset of central apnea with stepwise increase in ventilator rate

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Claure, Principal Investigator — University of Miami; Eduardo Bancalari, Principal Investigator — University of Miami; Deepak Jain, Principal Investigator — University of Miami
Locations (1):
- NICU at Holtz Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No